CLINICAL TRIAL: NCT07292376
Title: Implementing VTE Prevention in Ambulatory Cancer Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Karlyn Martin, Associate Professor of Medicine, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FP00005110
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Venous Thromboembolism; Neoplasms
MeSH Terms: conditions — Venous Thromboembolism; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical program (Other)
  Interventions: Other: Clinical program

INTERVENTIONS:
Other: Clinical program — Revised Vermont Model clinical program, including standardized education and training for oncology care team, clinical decision support and revised workflow for VTE risk assessment and thromboprophylaxis.

SUMMARY:
assess effectiveness of a , compared with usual care, to assess

The goal of this study is to learn if a modified clinical program can improve adherence to guideline recommendations for prevention of venous thromboembolism in ambulatory patients with cancer. The main question[s] it aims to answer are:

Does the modified program improve number of ambulatory oncology patients starting systemic treatment getting VTE risk-assessment? Does the modified program improve the number of patients receiving appropriate preventative anticoagulation? Researchers will compare to usual care (no clinical program).

Participant clinicians will be asked to

* receive education about VTE prevention recommendations
* carry out risk assessment, anticoagulation discussions, and document the results Participant patients will receive care from clinicians participating in the study as part of their cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians: practicing oncologist at study clinic site (UVMMC)
* Patients: diagnosis of cancer; starting new systemic cancer-directed therapy at a study clinic site under the direction of the enrolled clinician

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Documented VTE risk assessment | 30 days after new patient appointment
  Proportion of new patients who have documented VTE risk assessment

SECONDARY OUTCOMES:
Appropriate thromboprophylaxis | 30 days after new patient appointment
  Proportion of identified high-risk patients with prescription for thromboprophylaxis and low-risk patients without thromboprophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Karlyn Martin, MD, Principal Investigator — University of Vermont
Locations (1):
- Vermont Health, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No